CLINICAL TRIAL: NCT06913920
Title: A Two-Arm, Single-Blinded Randomized Controlled Trial Evaluating the Effectiveness of Mechanical Modalities Combined With Standard Therapy Versus Standard Therapy Alone for Edema and Pain Management After Distal Radius Fracture Fixation
Brief Title: Mechanical Modalities vs. Standard Care for Edema and Pain Management After DRF Fixation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al Hayah University In Cairo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMDRF2025-02
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Distal Radius Fractures
MeSH Terms: conditions — Wrist Fractures | interventions — Motion Therapy, Continuous Passive; Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two parallel arms. The Mechanical Modality Group (MMG) receives both mechanical devices (CPM and IPC) integrated with standard therapy. The Standard Care Group (SCG) receives the same standard therapy without the addition of mechanical modalities.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical Modality Group (MMG) (Experimental): Participants in the MMG will undergo a combined intervention that utilizes mechanical modalities in addition to a standard rehabilitation program.
  Interventions: Device: Continuous Passive Motion (CPM); Device: Intermittent Pneumatic Compression (IPC); Behavioral: Standard Therapy Program
- Standard Care Group (SCG) (Active Comparator): Participants in the SCG will receive the standard rehabilitation program alone without the application of mechanical devices.
  Interventions: Behavioral: Standard Therapy Program

INTERVENTIONS:
Device: Continuous Passive Motion (CPM) — Materials: A CPM device configured for wrist flexion-extension with an adjustable range of motion set between 0° and 30°.
  Procedure:
  The participant's wrist is gently secured in the device. The CPM device is programmed to deliver 20 minutes of continuous, passive motion through the set range.
  Device settings (e.g., speed) may be modified if the participant reports pain >4/10 on the NPRS.
  Arms: Mechanical Modality Group (MMG)
Device: Intermittent Pneumatic Compression (IPC) — Materials: An IPC sleeve designed for the forearm-to-hand region with a baseline compression setting of approximately 30 mmHg.
  Procedure:
  After CPM treatment, the IPC device is applied to the affected limb. The sleeve provides 15 minutes of intermittent compression with programmed intervals of inflation and deflation.
  Compression levels may be adjusted based on participant comfort and pain ratings.
  Arms: Mechanical Modality Group (MMG)
Behavioral: Standard Therapy Program — Procedures:
  Active/active-assisted wrist/forearm range of motion exercises led by a certified hand/physical therapist.
  Progressive grip-strengthening exercises using resistance bands or putty. Manual edema management techniques, including gentle massage and manual lymphatic drainage, as well as scar mobilization if needed.

SUMMARY:
This single-blinded, randomized controlled trial (RCT) will evaluate the added benefit of mechanical modalities (continuous passive motion (CPM) and intermittent pneumatic compression (IPC)) when integrated into standard therapy for managing postoperative edema and pain in patients undergoing distal radius fracture (DRF) fixation. The primary outcomes are edema volume (measured via volumeter) and pain intensity (Numeric Pain Rating Scale, NPRS) at 6 weeks post-operation. Secondary outcomes include wrist/forearm range of motion (ROM), grip strength, Patient-Rated Wrist Evaluation (PRWE), and adverse events.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years or older. Undergoing surgical treatment for distal radius fracture with stable internal fixation.

Able to initiate formal rehabilitation approximately 2 weeks postoperatively. Willing and able to attend in-clinic therapy sessions at the outpatient hand therapy center.

Exclusion Criteria:

Unstable fixation or need for further surgical intervention. Pre-existing conditions that would significantly affect upper limb function (e.g., severe arthritis, neurological disorders).

History of skin conditions or allergies that contraindicate the use of mechanical devices.

Any contraindication to mechanical modalities (for example, severe peripheral vascular disease).

Inability to comply with study procedures or follow-up visits. Pregnant or breastfeeding individuals.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Edema Volume | Assessed at baseline (2 weeks postoperatively) and at 6 weeks post-operation.
  Edema of the wrist/forearm will be quantitatively measured using a volumeter method. Lower volumes are indicative of reduced swelling.
Pain Intensity | Assessed at baseline (2 weeks postoperatively) and at 6 weeks post-operation.
  Pain is measured using the Numeric Pain Rating Scale (NPRS), with scores ranging from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Wrist/Forearm Range of Motion (ROM) | Measured at baseline, 6 weeks, and 3 months postoperatively.
  Active ROM is measured using a standard goniometer. Improvements in ROM indicate better recovery of function.
Grip Strength | Assessed at baseline, 6 weeks, and 3 months postoperatively.
  Evaluated using a calibrated dynamometer. Increased grip strength is suggestive of improved functional recovery.
Incidence of Adverse Events | Continuously monitored from baseline to the 3-month follow-up.
  All adverse events, including skin irritation or device intolerance, will be monitored and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Al Hayah University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No